CLINICAL TRIAL: NCT00265707
Title: A Study to Evaluate the Safety and Effectiveness (Overall Performance) of the Press-O-Sense Non-Invasive Blood Pressure Measuring Device.
Brief Title: Evaluation of a New Blood Pressure Measuring Device.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maaynei Hayesha Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DPTYN001CTIL
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2005-12

CONDITIONS: Hypertension
Keywords: Hypertension; Hypotension
MeSH Terms: conditions — Hypertension; Hypotension | interventions — Blood Pressure Determination

INTERVENTIONS:
Device: Blood pressure measurement

SUMMARY:
* A disposable blood pressure measuring device will be tested and compared to a standard mercury sphygmomanometer.
* Up to 100 subjects with various levels of blood pressure values will be tested.

DETAILED DESCRIPTION:
The study will comprise 85 to 100 subjects with blood pressure values ranging between 90 and 170mmHg -systolic and 65-95 -diastolic.

* Three sets of measurements will be performed on each subject. The measurement with the tested device placed between twh determinations with a mercury sphygmomanometer.
* Each measurement will be performed simultaneously by two examiners specially trained.
* Informed consent will be obtained from all participants.
* The results will be evaluated by a standard statistical plan ANSI/AAMI SP-10 2002.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or above
* Signed written informed consent

Exclusion Criteria:

* A history of cardiac arrythmia
* Wrist circumference smaller than 13cm or larger than 19.5cm
* Documented peripheral vascular disease
* Damage or injury to the left wrist
* Participation in any other clinical study
* Any acute coronary of cardiovascular illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09; Study Completion 2005-12

PRIMARY OUTCOMES:
The difference between the paired measurements with the tested device and the reference measurements (with a mercury sphygmomanometer) will differ by no more than +-5mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Mordchai Ravid, MD FACP, Principal Investigator — Maaynei Hayesha Hospital
Locations (1):
- Department of Medicine, Maaynei Hayesha Hospital, Tel Aviv, Israel